CLINICAL TRIAL: NCT00939549
Title: Phase II Study of High Dose Cyclophosphamide Followed by Glatiramer Acetate in the Treatment of Relapsing Remitting Multiple Sclerosis
Brief Title: High Dose Cyclophosphamide Followed by Glatiramer Acetate in the Treatment of Relapsing Remitting Multiple Sclerosis
Acronym: HiCy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study revised to retrospective chart review
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00016884
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: High dose cyclophosphamide
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Cyclophosphamide; Glatiramer Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High-dose cyclohosphamide (Experimental)
  Interventions: Drug: Cyclophosphamide/Glatiramer acetate

INTERVENTIONS:
Drug: Cyclophosphamide/Glatiramer acetate — Cyclophosphamide 50 mg/kg IV each day for four consecutive days. Glatiramer acetate 20 mg SC daily for 1 year.

SUMMARY:
The purpose of this study is to determine if high-dose cyclophosphamide followed by a maintenance dose of glatiramer acetate is safe in patients with relapsing remitting multiple sclerosis (MS). The investigators hypothesize that institution of glatiramer acetate treatment following high-dose cyclophosphamide treatment will extend the period of disease free activity and further reduce the disability in patients with relapsing remitting multiple sclerosis. The investigators plan to investigate the properties of glatiramer acetate against the recurrence of MS disease activity following high dose cyclophosphamide induced cessation detectable autoimmunity. The investigators hypothesize that glatiramer acetate, given in the phase of immune reconstitution after high-dose cyclophosphamide, may bias the immune system to a more tolerated state, thus leading to more stable and potentially permanent remissions.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an autoimmune disease characterized by progressive immune-mediated destruction of myelin and axons within the CNS. Despite the development, approval and clinical utilization of several medicines for patients with MS, most patients continue to accrue progressive disability. High-dose cyclophosphamide is chemotherapy treatment option for severe, refractory, immune-mediated illnesses such as MS. There is growing evidence that high dose cyclophosphamide is well tolerated and effective in MS. Our experience with 9 patients who underwent treatment at the Johns Hopkins Hospital yielded impressive results with a significant 40% reduction in baseline disability and an 81% reduction in MRI gadolinium enhancing lesions. Five out of 9 patients had recurrence of new brain MRI lesions during 24 months of follow-up, recurring in 4 patients during the first year of follow-up. Our findings suggest that high-dose cyclophosphamide holds promise in inducing remission and reducing disability in relapsing remitting MS however the recurrence of MS disease activity (evidenced by worsening disability, clinical exacerbations or ongoing MRI evidence of new lesions) suggests that high-dose cyclophosphamide given as a treatment on its own, is not sufficient to induce long-term remission.

Glatiramer acetate has been shown to be a more general suppressor of autoimmune disease, inhibiting the onset of experimental animal models of uveoretinitis, rheumatoid arthritis, immune rejection of grafts against host and host against graft disease, and inflammatory bowel disease. Glatiramer acetate was originally developed based on the observation that it inhibited the onset of clinical disease in an animal model of multiple sclerosis, experimental autoimmune encephalomyelitis (EAE). Glatiramer acetate suppression of EAE was found to be a general phenomenon not restricted to a particular species, disease type or encephalitogen used for the induction of EAE. A unique feature of glatiramer acetate is its promiscuous binding with high affinity to various class II MHC molecules and it potent induction of Th2 regulatory T cells. Moreover glatiramer acetate has subsequently been shown to be a more general suppressor of autoimmune disease, inhibiting the onset of experimental uveoretinitis, immune rejection of grafts against host and host against graft disease, and experimental inflammatory bowel disease.

We plan to investigate the properties of glatiramer acetate against the recurrence of MS disease activity following high dose cyclophosphamide induced cessation detectable autoimmunity. This study is a prospective, open-label two-year follow-up study in 12 patients with relapsing-remitting MS who are unable to tolerate or have failed to optimally respond to conventional therapy and are at high risk of disease progression and loss of function. Patients who elect to enter the study will be given a single course of high-dose, cyclophosphamide regimen without transplantation. Patients will then receive 20 mg of glatiramer acetate subcutaneously 4 to 6 weeks after the last dose of high-dose cyclophosphamide, to allow the immune system to have time to begin to reconstitute without glatiramer acetate but still provide sufficient time for glatiramer acetate to vaccinate against recurrence of MS disease activity.

The primary outcome of this pilot study will be to determine if high followed by a maintenance dose of glatiramer acetate is safe in this patient population. We hypothesize that institution of glatiramer acetate treatment following high-dose cyclophosphamide treatment will extend the period of disease free activity and further reduce the disability in patients with relapsing remitting MS.

ELIGIBILITY:
Inclusion criteria

1. Males and females between the ages of 18 and 70 years, inclusive.
2. Diagnosis of clinically definite MS according to the McDonald Criteria.
3. Must have been on conventional immunomodulatory treatment (interferon beta-1a, glatiramer acetate, or natalizumab) for at least 3 months OR have not tolerated conventional treatment OR have refused to start conventional treatment.
4. 2 or more total gadolinium enhancing lesions on each of two pretreatment MRI scans at screening and enrollment.
5. Subject must have EDSS ranging from 1.5 to 6.5.
6. Subject must have had at least one clinical exacerbation in the last year and this must have occurred after having been on Avonex, Betaseron, Copaxone, Rebif or Natalizumab therapy for at least 3 months. This does not apply if subject has refused to start conventional therapy.
7. Subject must have had a sustained (≥ 3 months) increase of > 1.0 on the EDSS (historical estimate allowed) between 3.0 and 5.5 or > 0.5 between 5.5 and 6.5 (while on therapy).
8. Written informed consent prior to any testing under this protocol, including screening tests and evaluations that are not considered part of the subject's routine care.
9. Women of childbearing potential should have a negative pregnancy test prior to entry into the study.

Exclusion criteria

1. Any risk of pregnancy--ALL female patients must have an effective means of birth control or be infertile due to hysterectomy, fallopian tube surgery, or premature menopause.
2. Cardiac ejection fraction of < 45%.
3. Serum creatinine > 2.0.
4. Patients who are pre-terminal or moribund.
5. Bilirubin > 2.0, transaminases > 2x normal.
6. Patients with EDSS < 3.0 or > 6.5.
7. Patients with pacemakers and implants who cannot get serial MRIs.
8. Patients with active infections until infection is resolved.
9. Patients with WBC count < 3000 cells/µl, platelets < 100,000 cells/µl and untransfused hemoglobin < 10 g/dl.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Safety - Serious adverse events | 2 years

SECONDARY OUTCOMES:
Radiologic - reduction in the number of gadolinium enhancing lesions, T2 plaque burden, and change in brain parenchymal fraction. | 2 years
Clinical/Neurological - Change in disability | 2 years
Immunological - change in immune profile | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Justin McArthur, MBBS, MPH, Principal Investigator — Johns Hopkins University; Robert Brodsky, M.D, Principal Investigator — Johns Hopkins University; Daniel Harrison, MD, Study Director — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital Multiple Sclerosis Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Krishnan C, Kaplin AI, Brodsky RA, Drachman DB, Jones RJ, Pham DL, Richert ND, Pardo CA, Yousem DM, Hammond E, Quigg M, Trecker C, McArthur JC, Nath A, Greenberg BM, Calabresi PA, Kerr DA. Reduction of disease activity and disability with high-dose cyclophosphamide in patients with aggressive multiple sclerosis. Arch Neurol. 2008 Aug;65(8):1044-51. doi: 10.1001/archneurol.65.8.noc80042. Epub 2008 Jun 9. PMID 18541787